CLINICAL TRIAL: NCT02056431
Title: Balancing Treatment Outcomes and Medication Burden Among Patients With Symptomatic Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CE-1304-7250
Record Dates: First submitted 2014-01-31; First posted 2014-02-06 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetes; Neuropathy; Patient-Reported Outcomes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVR Intervention Group (Experimental): Participants will receive 3 interactive voice response (IVR) calls (2nd, 4th, and 6th month post-treatment start date) to collect information on medication use, side effects, rating of side effects, and pain symptoms to be fed back to their physicians.
  Interventions: Behavioral: IVR Intervention Group
- IVR Control Group (No Intervention): Participants will receive 3 non-interactive voice response (IVR) calls (2nd, 4th, and 6th month post-treatment start date) containing general messages regarding diabetic education.

INTERVENTIONS:
Behavioral: IVR Intervention Group — Participants will receive 3 interactive voice response (IVR) calls (2nd, 4th, and 6th month post-treatment start date) to collect information on medication use, side effects, rating of side effects, and pain symptoms to be fed back to their physicians.
  Arms: IVR Intervention Group

SUMMARY:
Painful diabetic peripheral neuropathy (DPN) affects more than 5.5 million people with diabetes. People with painful DPN have trouble sleeping, participating in social events, and conducting daily activities such as going to the store. Several prescription medications are available for the treatment of DPN symptoms, but none work perfectly and all have side effects that may be difficult for some patients.

When patients report their symptoms and side effects to their doctor, they provide the doctor with important information to help them make adjustments to treatment that will help with symptoms and that the patient can tolerate in terms of side effects. In some cases, doctors may encourage patients to make these changes on their own at home based on their experience with therapy. However, patients may have a long time between visits to their doctor and may have trouble describing their symptoms to their doctor during a brief 10 to 15 minute visit.

This clinical trial explores the possibility of computerized telephone calls to patients (Interactive Voice Response, IVR, technology) to gather information about treatment experiences that can then be reported to the doctor or used to guide patients to make changes in how they take the medication. It addresses the following question: Can routinely asking patients about their experiences with medications and using that information to encourage clinically appropriate titration improve patient quality of life?

The investigators hypothesize that systematic collection and feedback of information about DPN treatment preferences and experience from newly treated patients to their primary care physician will facilitate treatment changes that improve patient outcomes

DETAILED DESCRIPTION:
Among newly-treated Diabetic Peripheral Neuropathy (DPN) patients, the investigators will compare the systematic collection and feedback of information about patients' treatment experiences on changes in quality of life (intervention group) to newly treated DPN patients in usual care who will receive generic educational messages by phone but no active data collection and feedback (comparator group). The investigators have chosen usual care as the control to evaluate the potential for the intervention to enhance current practice.

Aim 1: Refine and pilot test instruments for collecting the patient-reported data most important for guiding changes in treatment.

Aim 2: Implement a seven-month cluster randomized trial to improve quality of life among patients newly treated for DPN symptoms by collecting data on patient treatment experiences and facilitating evidence-based patient and provider-initiated treatment titration.

Aim 3: Examine patient and physician initiated treatment changes as secondary outcomes in order to inform the development of this type of rapid feedback process for guiding decision making about initial treatment selection among patients with DPN.

ELIGIBILITY:
Inclusion Criteria:

* All patients newly prescribed medication to treat diabetic peripheral neuropathy symptoms.

Exclusion Criteria:

* Patients with any evidence of use of diabetic peripheral neuropathy study medications.
* Patients with evidence of gestational diabetes (ICD-9: 648.8) due to variation in treatment and monitoring for women who are pregnant.
* Patients who simultaneously received a new diagnosis for depression or seizure conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1270 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyce S. Adams, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Division of Research Kaiser Permanente, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adams AS, Bayliss EA, Schmittdiel JA, Altschuler A, Dyer W, Neugebauer R, Jaffe M, Young JD, Kim E, Grant RW; Diabetes Telephone Study Team. The Diabetes Telephone Study: Design and challenges of a pragmatic cluster randomized trial to improve diabetic peripheral neuropathy treatment. Clin Trials. 2016 Jun;13(3):286-93. doi: 10.1177/1740774516631530. Epub 2016 Mar 31. PMID 27034455
- [Derived] Adams AS, Schmittdiel JA, Altschuler A, Bayliss EA, Neugebauer R, Ma L, Dyer W, Clark J, Cook B, Willyoung D, Jaffe M, Young JD, Kim E, Boggs JM, Prosser LA, Wittenberg E, Callaghan B, Shainline M, Hippler RM, Grant RW. Automated symptom and treatment side effect monitoring for improved quality of life among adults with diabetic peripheral neuropathy in primary care: a pragmatic, cluster, randomized, controlled trial. Diabet Med. 2019 Jan;36(1):52-61. doi: 10.1111/dme.13840. Epub 2018 Nov 7. PMID 30343489

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IVR Intervention Group | IVR Control Group
Started | 604 | 666
Completed | 560 | 619
Not Completed | 44 | 47

BASELINE CHARACTERISTICS:
Groups:
- IVR Intervention Group: Participants will receive 3 interactive voice response (IVR) calls (2nd, 4th, and 6th month post-treatment start date) to collect information on medication use, side effects, rating of side effects, and pain symptoms to be fed back to their physicians.
  IVR Intervention Group: 595 participants will receive 3 interactive voice response (IVR) calls (2nd, 4th, and 6th month post-treatment start date) to collect information on medication use, side effects, rating of side effects, and pain symptoms to be fed back to their physicians.
- Total: Total of all reporting groups
Arm/Group | IVR Intervention Group | IVR Control Group | Total
Number analyzed (Participants) | 604 | 666 | 1270
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (12.0) | 67.0 (11.5) | 67.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 329 | 349 | 678
  Male | 275 | 317 | 592
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 1 | 1 | 2
  Asian | 54 | 50 | 104
  Native Hawaiian or Pacific Islander | 2 | 7 | 9
  Black or African American | 79 | 88 | 167
  White | 343 | 375 | 718
  More than One Race | 3 | 4 | 7
  Hispanic | 115 | 133 | 248
  Unknown | 7 | 8 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 604 | 666 | 1270

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Quality of Life at Baseline and 8 Months
Description: The primary outcome measure is change in quality of life from baseline at eight months following study entry. We calculated the EuroQOL (EQ-5D) from the Global Health Scale, a 10-item Patient-Reported Outcomes Measurement Information System measure developed and validated in patients with neuropathy as part of the Quality of Life in Neurological Disorders Measures. The range for EQ-5D is 0-1, with "0" being the worst and "1" being the best.
Time Frame: Baseline and 8 months
Population: 1179 patients completed the close out survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IVR Intervention Group | IVR Control Group
Number analyzed (Participants) | 561 | 618
units on a scale
  Baseline time-point | 0.66 (0.10) | 0.65 (0.10)
  8 Month time-point | 0.68 (0.10) | 0.68 (0.10)

2. Secondary Outcome: Number of Participants With Minimally Effective Dose in 12 Months
Description: Count of patients who ever received a minimally effective dose of the medications they started on during the 12 months following treatment start (measured post only).
Time Frame: 12 months
Population: 1179 Patient completed the close out survey
Measure: Count of Participants; unit: Participants
Groups:
- IVR Control Group: Participants will receive 3 non-interactive voice response (IVR) calls (2nd, 4th,and 6th months post start date) containing generic messages regarding diabetes education
- IVR Intervention Group: Participants will receive 3 interactive voice response (IVR) calls (2nd, 4th,and 6th months post start date) to collect information on medication use, side effects, rating of side effects and pain symptoms to be fed back to their physicians
Arm/Group | IVR Control Group | IVR Intervention Group
Number analyzed (Participants) | 618 | 561
Participants | 299 | 290

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant from the time of enrollment through 8 months.
Description: Given that this is a low risk study, we do not anticipate that any of the adverse events are associated with the intervention itself. We created an algorithm to extract information on deaths among participants from the electronic medical record every 6 months and reported these to the independent safety monitor.
Arm/Group | IVR Intervention Group | IVR Control Group
Serious Adverse Events (participants affected / at risk) | 138/604 | 149/666
Other Adverse Events (participants affected / at risk) | 0/604 | 0/666
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVR Intervention Group (N=604) | IVR Control Group (N=666)
Death (General disorders) | 20 (20) | 24 (24) — We created an algorithm to extract information on all hospitalizations and deaths in our population regardless of organ system.
Any Hospitalizations Occurring During the Study Period (General disorders) | 118 (118) | 125 (125) — We did not collect cause of death due to a 2-year lag between the time of death and assignment of the cause of death by the state.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No